BD1412-62CEC Bioequivalence and secondarily drug-drug interaction of fixed combination of Metformin/Gliclazide fixed compared with the co-administrarion of individual tablets EMR200763-003 Version 1.0

#### Statistical Analysis Plan

**Clinical Trial Protocol** Identification No.

BD1412-62CEC EMR200763-003

Title:

Randomized, Open label, Single Dose, 4-treatments, 4-periods, Crossover design (4 x 4) Study to evaluate the Bioequivalence and Secondarily Drug - Drug Interaction of Fixed Combination of Metformin Tablets 1000 mg/Gliclazide 30 mg MR, Compared with the Co-administration of Individual Tablets and Individual Administration of Each single tablet (Metformin 1000 mg XR and Gliclazide 30 mg MR) in Healthy Volunteers.

**Trial Phase** T

**Investigational Medicinal** Product(s)

Metformin/Gliclazide

**Clinical Trial Protocol** Version

2 October 2017/Version 1.0

Statistical Analysis Plan

Author

Agust 2018/Version 1.0

PPD

Statistical Analysis Plan **Date and Version** 

Statistical Analysis Plan

Reviewers



This document is the property of Merck KGaA, Darmstadt, Germany, or one of its

It is intended for restricted use only and may not - in full or part - be passed on, reproduced, published or used without express permission of Merck KGaA, Darmstadt, Germany or its affiliate.

Copyright © 2017 by Merck KGaA, Darmstadt, Germany or its affiliate. All rights reserved.

#### 1. Signature Page

Statistical Analysis Plan: BD1412-62CEC EMR200763-003

Randomized, Open label, Single Dose, 4-treatments, 4-periods, Crossover design (4 x 4) Study to evaluate the Bioequivalence and Secondarily Drug - Drug Interaction of Fixed Combination of Metformin Tablets 1000 mg/Gliclazide 30 mg MR, Compared with the Coadministration of Individual Tablets and Individual Administration of Each single tablet (Metformin 1000 mg XR and Gliclazide 30 mg MR) in Healthy Volunteers.



# 2. Table of Contents

| 1 | | Singature page | 2 |
|---|---|---|---|
| 2 | | Table of contents | 3 |
| 3 | | List of abbreviation and definition of terms | 4 |
| 4 | | Modification history | 6 |
| 5 | | Purpose of the statistical analysis plan | 6 |
| 6 | | Summary of clinical trial features | 6 |
| | 6.1 | Primary objectives and endpoint | 6 |
| | 6.2 | Secondary objectives and endpoint | 7 |
| | 6.3 | Overall trial design and plan | 7 |
| 7 | | Sample size | 8 |
| 8 | | Overview of planned analyses | 9 |
| | 8.1 | Interim analysis | 9 |
| 9 | | Changes to the planned analyses in the clinical trial protocol | 10 |
| 10 | | Protocol deviations and analysis sets | 10 |
| | 10.1 | Definition of protocol deviations and analysis sets | 10 |
| 11 | | General specifications of statistical analyses | 11 |
| 12 | | Protocol deviations | 11 |
| | 12.1 | Important protocol deviations | 11 |
| | 12.2 | Reasons leading to the exclusion from an analysis set | 11 |
| 13 | | Demographics and other baseline characteristics | 12 |
| | 13.1 | Demographics | 12 |
| 14 | | Treatment compliance and exposure | 13 |
| 15 | | Endpoint evaluation | 14 |
| | | Primary endpoint analyses | 14 |
| | 15.2 | Bioavailability statistics | 14 |
| | 15.3 | Box and whiskers plots | 17 |
| | 15.4 | Secondary endpoint analyses | 20 |
| | 15.5 | Other endpoint analyses | 22 |
| 16 | | Estimation of individual pharmacokinetic parameters | 32 |
| 17 | | Safety evaluation | 34 |
| | 17.1 | Pharmacokinetic parameter's outliers | 34 |
| 18 | | Averse events | 38 |
| 19 | | References | 38 |
| 20 | | Appendices | 38 |

3

#### List of Abbreviations and Definition of Terms

AE Adverse Event

AUC Area under the plasma concentration-time curve

AUC $_{0\rightarrow\infty}$  The AUC from time zero (dosing time) extrapolated to infinity

AUC<sub>0 $\rightarrow$ t</sub> The AUC from time zero (= dosing time) to the last sampling time (t<sub>last</sub>) at

which the concentration is at or above the lower limit of quantification

AUCextra% The AUC from time t<sub>last</sub> extrapolated to infinity given as percentage of

 $AUC_{0\rightarrow\square}$ 

BE Bioequivalence

BMI Body Mass Index

CI Confidence Interval

CL/f The apparent total body clearance of drug following extravascular

administration.

C<sub>max</sub> Maximum observed plasma concentration

CRF Case Report Form

CRO Contract Research Organization

CSR Clinical Study Report
CTR Clinical Trial Report

CTMS Clinical Trial Management System

CTP Clinical Trial Protocol

CV Coefficient of Variation (%)

CYP Cytochrome P 450 ECG Electrocardiogram

ECOG Eastern Cooperative Oncology Group

eCRF Electronic Case Report Form

GCP Good Clinical Practice

GeoCV% Geometric Coefficient of Variation

GeoMean Geometric Mean

GIR Glucophage Immediate Release

HR Hazard ratio

# BD1412-62CEC Bioavailability of a Metformin/Gliclazide fixed combination tablet Version 1.0

HAV Hepatitis A Virus

HbA<sub>1C</sub> Glycosylated Hemoglobin Type A<sub>1C</sub>

HBsAg Hepatitis B Surface Antigen

HCV Hepatitis C Virus

HIV Human Immunodeficiency Virus

ICF Informed Consent Form

ICH International Conference on Harmonization

IMP Investigational Medicinal Product

LLOQ Lower Level of Quantification

Max Maximum

Mean Arithmetic mean

Min Minimum

MedDRA Medical Dictionary For Regulatory Activities

MRI Magnetic Resonance Imaging
MSS Merck Santé s.a.s. in Semoy

N Number of non-missing observations

PK Pharmacokinetics
PR Partial Response
PT Preferred team
OoL Quality of Life

SAE Serious Adverse Event

SASS Sino-American Shanghai Squibb Pharmaceuticals Ltd

SAP Statistical Analysis Plan SBP Systolic Blood Pressure

SD Standard Deviation

SDTM Study Data Tabulation Model

SEM Standard Error of the Mean

SOC System Organ Class

t1/2 Apparent terminal half-lifeT2DM Type 2 Diabetes Mellitus

TEAE Treatment-Emergent Adverse Event

TLF Tables, Listings, and Figures

| BD1412-62CEC<br>EMR200763-003 | Bioavailability of a Metformin/Gliclazide fixed combination tablet Version 1.0 |
|---|---|
| tlast | The last sampling time at which the concentration is at or above the lower limit of quantification |
| $t_{ m max}$ | The time to reach the maximum observed concentration |
| TP | Treponema Pallidum |
| $V_{z/f}$ | Apparent volume of distribution during the terminal phase following extravascular administration |
| $\lambda_z$ | Terminal elimination rate constant |
| WHO | World Health Organisation |

# 4 Modification History

| Unique<br>Identifier for<br>SAP Version | DATE OF SAP<br>Version | Author | CHANGE DESCRIPTION from the previous version | LEVEL |
|---|---|---|---|---|
| | March 2019 | PPD | New Document | 1.0 |

# 5 Purpose of the Statistical Analysis Plan

The purpose of this SAP is to document technical and detailed specifications for the final analysis of data collected for protocol BD1412-62CEC EMR200763-003. Results of the analyses described in this SAP will be included in the Clinical Study Report (CSR). Additionally, the planned analyses identified in this SAP will be included in regulatory submissions or future manuscripts. Any post-hoc.

The SAP is based upon section 9 (Statistical and Pharmacokinetical Analysis) of the trial protocol and is prepared in compliance with ICH E9.

# 6 Summary of Clinical Trial Features

#### 6.1 Primary Objectives and Endpoints

- To demonstrate bioequivalence of the fixed combination of Metformin tablets 1000 mg XR plus Gliclazide 30 mg MR compared to the co-administration of the individual tablets of Metformin 1000 mg XR and Gliclazide 30 mg MR, given as single dose to healthy volunteers in fasting state. Primary endpoints will be AUC0-t, AUC0-∞ and Cmax for Metformin and Gliclazide.
- To demonstrate the lack of an effect of Gliclazide on the PK of Metformin by comparing the Metformin PK following administration of the fixed combination tablet Metformin/Gliclazide and Metformin alone (AUC0-t, AUC0-∞ and Cmax of Metformin).
- To demonstrate the absence of an effect of Metformin on the PK of Gliclazide by comparing the Gliclazide PK following administration of the fixed combination tablet Metformin/Gliclazide and Gliclazide alone (AUC0-t, AUC0-∞ and Cmax of Gliclazide).

# 6.2 Secondary Objectives and Endpoints

- The secondary endpoints variable are volume of distribution Ke, half-life elimination, clearance, and median residence time all these parameters will be presented only for informative reasons for both medications.
- To compare the safety and tolerability of all the experimental treatments.

#### 6.3 Overall Trial Design and Plan

This randomized, open-label, single dose, four-treatment, four period crossover design (4x4) trial with a 14-day wash-out period along 4 study stages will investigate the bioequivalence (primary endpoints are AUC0-t, AUC0-∞ or Cmax for Metformin and Gliclazide) of a Metformin/Gliclazide fixed combination tablet (1000 mg /30 mg MR) compared with the co-administration of the individual tablets (Metformin 1000 mg and Gliclazide 30 mg MR) and the drug-drug interaction between the Metformin/Gliclazide fixed combination and the administration of each single tablet, administered in fasted condition in 40 healthy volunteers. Secondarily, safety and tolerability will be also investigated in every case.

The subjects will be randomized to one of the 4 treatment sequences (see table below). Ten subjects will be randomized to each treatment sequence with a minimum proportion of 30% for each sex in each treatment sequence.

| Sequence | Period 1 | | Period 2 | | Period 3 | | Period 4 |
|---|---|---|---|---|---|---|---|
| 1 | Fixed combination | po | Metformin +<br>Gliclazide | po | Metformin | po | Gliclazide |
| 2 | Metformin +<br>Gliclazide | out period | Gliclazide | ut period | Fixed combination | ut period | Metformin |
| 3 | Metformin | Wash-0 | Fixed combination | Wash-0 | Gliclazide | Wash-0 | Metformin +<br>Gliclazide |
| 4 | Gliclazide | | Metformin | | Metformin +<br>Gliclazide | | Fixed combination |

# 7 Sample Size

The sample size estimation is based on the CV intrasubject variability of both drugs. Because the pharmacokinetic and drug-drug interaction, evaluates changes in the bioavailability, the propose is the use the same determination for both aims.

The sample size is determined by the primary endpoint with the greatest variability under fasting conditions, AUC0-t of Metformin (CV=23%). Assuming a mean treatment ratio of 0.95, and aiming at a power of 90% for the individual test, alpha=0.05 one-sided, 32 evaluable subjects are sufficient to demonstrate bioequivalence in the first step. The same arguments can be applied to the second step: Test absence of an effect of Gliclazide on the PK of Metformin, whereas the power for the third test is close to 100% with 32 subjects, due to the low variability of Gliclazide PK. Therefore, the overall power is still greater than 80% with 32 evaluable subjects. Considering a drop-out rate of approximately 20%, 40 subjects should be randomized.

According to NOM-177-SSA1-2013, this sample determination was realized with Chow & Wang (2001) equation

$$n \ge \left[t_{(\alpha,2n-2)} + t_{(\beta,2n-2)}\right]^2 \cdot \left(\frac{CV_{intra}}{\ln 0.8 - \ln \theta}\right)^2$$

Where:

t(alfa, 2n-2) and t(beta, 2n-2) considered the error alfa and beta respectively

CVintra: intra subject variability for crossover (or replicate crossover) study.

Tetha: 0.95: the target ratio in average BA between the two formulations expressed in percentage of the average reference

0.8: the least statistical power to detect (1-Power) differences between the Test and the Reference formulation (in this case the power expected is 90%)

# 8 Overview of Planned Analyses

Statistical analysis and analysis of PK parameters will be performed using Phoenix WinNonlin software Version 6.3 (PPD).

Descriptive statistical methods will be used to summarize demographic characteristics, pharmacokinetics parameters and adverse events. After the data base closing

Individual plasma concentration-time will be tabulated and plotted. Primary pharmacokinetics parameters, AUC and Cmax, will be tabulated and plotted by subject. Likewise, differences and odd ratios for test/reference will be tabulated for each subject for those parameters. Plasma concentration - time graphs will be made using arithmetic and semi-logarithmic scale. All de calculations will be determinated in concordance with NOM-177-SSA1-2013

The following sequential testing of a priori ordered hypotheses will be applied, as shown below. Bioequivalence test methodology will be used in all 3 steps:

- 1. Test bioequivalence of fixed combination and separate tablets
- 2. Test absence of an effect of Gliclazide on the PK of Metformin
- 3. Test absence of an effect of Metformin on the PK of Gliclazide

#### 8.1 Interim Analysis

Bioequivalence in step1:

A mixed model will be applied to log-transformed Cmax, AUC0-t and AUC0-∞ (both analytes) with treatment, period and sequence as fixed effects, and subject (sequence) as a random effect. Based on the residual error term 90% confidence intervals will be computed for the estimated

differences Test – Reference, resulting in 90% confidence intervals for the Test/Reference ratios after back-transformation.

Drug-drug interaction in steps 2 and 3:

A mixed model will be applied to log-transformed Cmax, AUC0-t and AUC0- $\infty$  (one analyte) with treatment as fixed effect, and subject as a random effect. Based on the residual error term 90% confidence intervals will be computed for the estimated differences Test – Reference, resulting in 90% confidence intervals for the Test/Reference ratios after back-transformation.

- 1. Bioequivalence will be concluded, if all six 90% CIs for all six primary endpoints reside within the acceptance range [0.80 1.25]
- 2. Absence of an effect of Gliclazide on the PK of Metformin will be concluded, if all three 90% CIs for Metformin endpoints reside within the range [0.80 1.25]
- 3. Absence of an effect of Metformin on the PK of Gliclazide will be concluded, if all three 90% CIs for Gliclazide endpoints reside within the range [0.80 1.25]

Additionally, the primary endpoints will be descriptively analyzed and graphical displays (Boxwhiskers-plots) will be prepared.

Statistical model in the variance analysis of mixed effects should be applied for log-transformed parameters Cmax, AUC0-t and AUC0-∞ (one analyte) with TREATMENT as fixed effect and SUBJECT as randomized effect. Based on residual errors, confidence interval of 90 % will be built for estimated differences for test - reference, resulting in a confidence interval of 90 % for the test/reference ratio following transformation.

Using minimum mean squares for AUC and Cmax, two-side t test will be performed (Schuirmann's test) by constructing confidence intervals of 90 % for test/reference ratios. If and only if intervals are within interval (80, 125), bioequivalence will be proven for both drugs.

Bioequivalence is concluded if 6 confidence intervals for the analytes are included into the bioequivalence limits.

#### 9 Changes to the Planned Analyses in the Clinical Trial Protocol

The statistical methods as described in the protocol were adopted.

There are no changes to the planned analyses.

#### 10 Protocol Deviations and Analysis Sets

# 10.1 Definition of Protocol Deviations and Analysis Sets

All deviations should be justified with statistical or scientific data and any change to the original statistical plan should be documented, in the study master file and in the pharmacokinetics statistical report as well as in the final study report. Subjects' data will not be replaced. Any missing

data will be considered as non-existent data. Likewise, data cannot be removed from the statistical analysis, except in the following events.

# Research Subjects with Pre-dose Concentrations in the Biological Matrix

In the event pre-dose concentration is < 5 % of the  $C_{max}$  value for a research subject, subject's data can be included without any adjustment to measurement and pharmacokinetic calculations. When pre-dose value is > 5 % of the  $C_{max}$ , research subject should be removed from all study bioequivalence assessments.

#### Exclusion of data due to vomit or diarrhea.

Data from research subjects who experience vomiting and diarrhea throughout the bioequivalence study for immediate release products can be removed from the statistical analysis if vomiting and diarrhea occur before 2 fold the median for  $t_{max}$  or 2 fold  $t_{max}$  value obtained from the research subject in a given period.

# Research subject with very low plasma concentrations for study drugs.

As established by NOM-177-SSA1-2013, research subjects in a cross designed who provide evaluable data for test drug and reference drug, or who do not have evaluable data in the single period of a parallel design, should not be either included in the statistical analysis.

It is considered that a research subject has very low concentrations, if the AUC is lower than 5 % of the geometric means for the reference drug's AUC (it should be calculated without including outliers). Exclusion of data due to this reason will only be accepted prior scientific rationale and review of the case by the COFEPRIS.

# 11 General Specifications for Statistical Analyses

Pharmacokinetic parameters (non-compartmental analysis) and statistical analysis for determining bioequivalence will be calculated using Phoenix WinNonlin 8.0 software.

The results of this trial will be reported using summary tables, figures, and data listings, as appropriate. All data will be summarized by treatment and/or scheduled time point, as appropriate.

#### 12 Protocol Deviations

# 12.1 Important Protocol Deviations

Not applicable. No deviation was observed in the study

# 12.2 Reasons Leading to the Exclusion from an Analysis Set

#### Research Subjects with Pre-dose Concentrations in the Biological Matrix

In the event pre-dose concentration is less than 5 % of the  $C_{max}$  value for a research subject, subject's data can be included. When pre-dose value is greater than 5 % of the  $C_{max}$ , research subjects data should be removed from all study of food effect on bioavailability.

#### Exclusion of data due to vomit or diarrhea.

Data from research subjects who experience vomiting and diarrhea throughout the study for immediate release products can be removed from the statistical analysis if vomiting and diarrhea occur before 2 fold the median for  $t_{max}$  or 2 fold  $t_{max}$  value obtained from the research subject in a given period.

#### Research subject with very low plasma concentrations for study drugs.

As established by NOM-177-SSA1-2013, research subjects in a cross designed who provide evaluable data for test drug and reference drug, or who do not have evaluable data in the single period of a parallel design, should not be either included in the statistical analysis.

It is considered that a research subject has very low concentrations, if the AUC is lower than 5 % of the geometric means for the reference drug's AUC (it should be calculated without including outliers). Exclusion of data due to this reason will only be accepted prior scientific rationale and review of the case by the COFEPRIS.

# 13 Demographics and Other Baseline Characteristics

Demographic data from each volunteer is shown in table 13.1 and the descriptive statistics for the demographic variables from volunteers recruited in the study are shown in table 13.2. PPD

# 13.1 Demographics

Table 13.1. Demographic Variables' Individual Data

| Case | Sex | Age | Weight | Height | BMI | Sequence |
|------|-----|-----|--------|--------|-----|----------|
| PPD | | | | | | |
| • | | | | | | |



Table 13.2. Demographic Variables' Descriptive Statistics

| Statistics | Age (years) | Weight (kg) | Height (m) | BMI<br>(Kg/m²) |
|------------|-------------|-------------|------------|----------------|
| Mean | PPD | | | |
| SD | | | | |
| Median | | | | |



#### 14 Treatment Compliance and Exposure

All subjects receive the investigational treatment at the pre-specified fixed dosage. Information relating to the extent of exposure is thus contained in the treatment labelling.

#### 15 Endpoint Evaluation

#### 15.1 Primary Endpoint Analyses

The determination of pharmacokinetics parameters were determined using WinNonlin software depending of their own characteristics as follows:

Cmax: is the peak or maximum concentration

AUC<sub>0-t</sub>: area under de curve computed from time zero to the time of the last positive Y value.

AUC<sub>0-∞</sub>: area under de curve computed from time zero to extrapolated from infinity.

Ke: First-order rate constant associated with the terminal (log-linear) elimination phase. This is estimated via linear regression of time vs. log concentration.

To demonstrate bioequivalence of the fixed combination of Metformin tablets 1000 mg XR plus Gliclazide 30 mg MR compared to the co-administration of the individual tablets of Metformin 1000 mg XR and Gliclazide 30 mg MR, given as single dose to healthy volunteers in fasting state. Primary endpoints will be AUC0-t, AUC0-∞ and Cmax for Metformin and Gliclazide.

To demonstrate the lack of an effect of Gliclazide on the PK of Metformin by comparing the Metformin PK following administration of the fixed combination tablet Metformin/Gliclazide and Metformin alone (AUC0-t, AUC0-∞ and Cmax of Metformin).

To demonstrate the absence of an effect of Metformin on the PK of Gliclazide by comparing the Gliclazide PK following administration of the fixed combination tablet Metformin/Gliclazide and Gliclazide alone (AUC0-t, AUC0-∞ and Cmax of Gliclazide).

#### 15.2 Bioavailability Statistics

In tables 15.2.1 and 15.2.2, pharmacokinetic equivalence statistical results are shown for the metformin's logarithmically transformed pharmacokinetic data, taking  $Dabex^{\mathbb{R}}XR + DiamicronMR^{\mathbb{R}}$  (B formulation) as reference drug. In tables 15.2.3 and 15.2.4, pharmacokinetic equivalence

statistical results are shown for the metformin's logarithmically transformed pharmacokinetic data, taking  $Dabex^{®}$  XR (C formulation) as the reference drug.

Table 15.2.1. Statistics for the Metformin's Pharmacokinetic Equivalence Determination. The Assessed Products are: Metformin-Gliclazide vs Dabex® XR + Diamicron MR®. (Dabex® XR as reference)

| D | Point | 90% Confidence | Two one te | D | |
|---|---|---|---|---|---|
| Parameter | Estimate | Interval | P < 80% | P > 125% | Power |
| LnC <sub>max</sub> | PPD | | | | |
| LnAUC <sub>0-t</sub> | | | | | |
| $LnAUC_{0-\infty}$ | | | | | |

Table 15.2.2. Statistics for the Metformin's Pharmacokinetic Equivalence Determination. The Assessed Products are: Metformin-Gliclazide vs Dabex<sup>®</sup> XR.

| Danamatan | Point | 90% Confidence | Two one te | Darran | |
|---|---|---|---|---|---|
| Parameter | Estimate | Interval | P < 80% | P > 125% | Power |
| LnC <sub>max</sub> | PPD | | | | |
| LnAUC <sub>0-t</sub> | | | | | |
| $LnAUC_{0-\infty}$ | | | | | |

Table 15.2.3. Statistics for the Metformin's Pharmacokinetic Equivalence Determination. The Assessed Products are: Dabex<sup>®</sup> XR vs Dabex<sup>®</sup> XR + Diamicron MR<sup>®</sup>. (Dabex<sup>®</sup> XR alone as reference)

| Damamatan | Point | 90% Confidence | Two one te | Dayyan | |
|---|---|---|---|---|---|
| Parameter | Estimate | Interval | P < 80% | P > 125% | Power |
| LnC <sub>max</sub> | PPD | | | | |
| LnAUC <sub>0-t</sub> | | | | | |
| LnAUC <sub>0-∞</sub> | | | | | |

Table 15.2.4. Statistics for the Gliclazide's Pharmacokinetic Equivalence Determination. The Assessed Products are: Metformin-Gliclazide vs Dabex® XR + Diamicron MR®. (Diamicron MR® as reference)

| Danamatan | Point | 90% Confidence | Two one | Darrag | |
|---|---|---|---|---|---|
| Parameter | Estimate | Interval | P < 80% | P > 125% | Power |
| LnC <sub>max</sub> | PPD | | | | |
| LnAUC <sub>0-t</sub> | | | | | |
| LnAUC <sub>0-∞</sub> | _ | | | | |

Table 15.2.5. Statistics for the Gliclazide's Pharmacokinetic Equivalence Determination. The Assessed Products are: Metformin-Gliclazide vs Diamicron MR<sup>®</sup>.

| Parameter | Point | 90% Confidence | Two one | Power | |
|---|---|---|---|---|---|
| Farameter | Estimate | Interval | P < 80% | P > 125% | Power |
| LnC <sub>max</sub> | PPD | | | | |
| LnAUC <sub>0-t</sub> | | | | | |
| $LnAUC_{0-\infty}$ | | | | | |

Table 15.2.6. Statistics for the Gliclazide's Pharmacokinetic Equivalence Determination. The Assessed Products are: Diamicron MR® vs Dabex® XR + Diamicron MR®. (Diamicron MR® alone as reference)

| Parameter | Point<br>Estimate | 90% Confidence<br>Interval | Two one te | Power | |
|---|---|---|---|---|---|
| | | | P < 80% | P > 125% | 1 |
| LnC <sub>max</sub> | PPD | | | | |
| LnAUC <sub>0-t</sub> | | | | | |
| LnAUC <sub>0-∞</sub> | | | | | |

As set for in the Mexican Official Standard, NOM-177-SSA1-2013, the parameters to be assessed in this study to establish the conclusion about the potential bioequivalence of drugs are  $C_{max}$  as indicative of the rate of absorption and the AUC as indicative of the absorbed amount. Results of bio-inequivalence are shown. PPD

Table 15.2.1 shows the results of the evaluation of the metformin and gliclazide given concomitantly versus the test formulation containing both drugs. PPD

In table 15.2.3, when the metformin reference drug is administered versus the concomitant administration of the reference drugs (metformin + gliclazide), appl

Tables 15.2.4, 15.2.5, and 15.2.6 show the gliclazide's pharmacokinetic equivalence results in all assessments made; PPD

The estimated statistical power was greater than 80 % for all the parameters assessed, which implies a good certainty to determine a bioequivalence and that the sample size was appropriate.

# PPD

#### 15.3 Box and Whiskers plots.

In tables 15.3.1 and 15.3.2, box and whiskers plots corresponding to the parameters used to assess the absorption and bioavailability for metformin and gliclazide, respectively, are shown.

| | Figure 15.3.1 Box and Whiskers Plot for the Metformin's Pharmacokinetic Parameters |
|---|---|
| PPD | |
| PPD | |

| | Table 15.3.2. Box and Whiskers Plot for the Gliclazide's Pharmacokinetic Parameters |
|---|---|
| PPD | |
| PPD | |

# 15.4 Secondary Endpoint Analyses

Average results of the metformin's pharmacokinetic parameters are shown in tables 15.4.1 for test formulation, 15.4.2 for metformin + gliclazide reference formulations and 15.4.3 for metformin reference. In these tables are shown the pharmacokinetics parameters determined for metformin.

Table 15.4.1. Metformin's Pharmacokinetic Parameters Results for test formulation

| | | | | | Metformin-Glid | clazide | | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | N | Mean | SD | CV% | Min | Max | Median | Geometric<br>Mean | CV% Geometric<br>Mean |
| AUC_%Extrap_obs | PPD | | | | | | | | |
| AUCINF_obs | | | | | | | | | |
| AUClast | | | | | | | | | |
| Cl_F_pred | | | | | | | | | |
| Cmax | | | | | | | | | |
| HL_Lambda_z | | | | | | | | | |
| MRTINF_obs | | | | | | | | | |
| Tmax | | | | | | | | | |
| Vz_F_pred | | | | | | | | | |

Table 15.4.2. Metformin's Pharmacokinetic Parameters Results for concomitant reference administration

| | | | | [ | abex® XR + Diam | icron MR® | | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | N | Mean | SD | CV% | Min | Max | Median | Geometric | CV% Geometric |
| | | | 30 | C V 76 | IVIIII | IVIAX | Median | Mean | Mean |
| AUC_%Extrap_obs | PPD | | | | | | | | |
| AUCINF_obs | | | | | | | | | |
| AUClast | | | | | | | | | |
| Cl_F_pred | | | | | | | | | |
| Cmax | | | | | | | | | |
| HL_Lambda_z | | | | | | | | | |
| MRTINF_obs | | | | | | | | | |
| Tmax | | | | | | | | | |
| Vz_F_pred | | | | | | | | | |

Table 15.4.3. Metformin's Pharmacokinetic Parameters Results for reference administration alone

| | | | | | Dabex® X | IR . | | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | N | Mean | SD | CV% | Min | Max | Median | Geometric<br>Mean | CV% Geometric<br>Mean |
| AUC_%Extrap_obs | PPD | | | | | | | | |
| AUCINF_obs | | | | | | | | | |
| AUClast | | | | | | | | | |
| Cl_F_pred | | | | | | | | | |
| Cmax | | | | | | | | | |
| HL_Lambda_z | | | | | | | | | |
| MRTINF_obs | | | | | | | | | |
| Tmax | | | | | | | | | |
| Vz_F_pred | | | | | | | | | |

Average results of the gliclazide's pharmacokinetic parameters are shown in tables 15.4.4 for test formulation, 15.4.5 for metformin + gliclazide reference formulations and 15.4.6 for gliclazide reference. In these tables are shown the pharmacokinetics parameters determined for metformin.

Table 15.4.4. Gliclazide's Pharmacokinetic Parameters Results for test formulation

| | | | | | Metformin-Gli | clazide | | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | N | Mean | SD | CV% | Min | Median | Max | Geometric Mean | CV% Geometric |
| | | | 30 | CV/6 | IVIIII | Median | IVIAX | Geometric Mean | Mean |
| AUC_%Extrap_obs | PPD | | | | | | | | |
| AUCINF_obs | | | | | | | | | |
| AUClast | | | | | | | | | |
| Cl_F_pred | | | | | | | | | |
| Cmax | | | | | | | | | |
| HL_Lambda_z | | | | | | | | | |
| MRTINF_obs | | | | | | | | | |
| Tmax | | | | | | | | | |
| Vz_F_pred | | | | | | | | | |

Table 15.4.5. Glicalzide's Pharmacokinetic Parameters Results for concomitant reference administration

| | | | | | Dabex® XR + Diam | icron MR® | | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | N | Mean | SD | CV% | Min | Median | Max | Geometric Mean | CV% Geometric<br>Mean |
| AUC_%Extrap_obs | PPD | | | | | | | | |
| AUCINF_obs | | | | | | | | | |
| AUClast | | | | | | | | | |
| Cl_F_pred | | | | | | | | | |
| Cmax | | | | | | | | | |
| HL_Lambda_z | | | | | | | | | |
| MRTINF_obs | | | | | | | | | |
| Tmax | | | | | | | | | |
| Vz_F_pred | | | | | | | | | |

Table 15.4.6. Gliclazide's Pharmacokinetic Parameters Results for reference administration alone

| | | | | | Diamicron N | MR® | | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | N | Mean | SD | CV% | Min | Median | Max | Geometric Mean | CV% Geometric |
| | | | 30 | CV /0 | IVIIII | iviculati | IVIAX | Geometric Mean | Mean |
| AUC_%Extrap_obs | PPD | | | | | | | | |
| AUCINF_obs | | | | | | | | | |
| AUClast | | | | | | | | | |
| Cl_F_pred | | | | | | | | | |
| Cmax | | | | | | | | | |
| HL_Lambda_z | | | | | | | | | |
| MRTINF_obs | | | | | | | | | |
| Tmax | | | | | | | | | |
| Vz_F_pred | | | | | | | | | |

# 15.5 Other Endpoint Analyses

Data about plasma concentration versus time for each subject, as well as the descriptive statistics are shown in tables 15.5.1 for metformin test formulation, 15.5.2 for metformin + gliclazide reference formulations concomitant administration and 15.5.3 for metformin reference alone administration.

Table 15.5.1. Individual concentrations table corresponding to metformin-gliclazide test formulation. n = P volunteers

| _ | Time | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Form | Volunteer | 0.0000 | 0.5000 | 1.0000 | 2.0000 | 3.0000 | 4.0000 | 5.0000 | 6.0000 | 7.0000 | 8.0000 | | | 16.0000 | 24.0000 | 28.0000 | 32.0000 | 48.0000 | 72.0000 | 96.0000 | 120.0000 | 144.0000 1 | 168.0000 |
| PPD | | 0.0000 | 0.0000 | 2.0000 | 2.0000 | 0.0000 | | 0.0000 | 0.0000 | 710000 | 0.0000 | 20,0000 | 22.0000 | 2010000 | 20000 | 20,000 | 02.0000 | 1010000 | 72.0000 | 50.000 | 220.0000 | | 200,0000 |

Table 15.5.2 Individual concentrations table for metformin + gliclazide, reference formulation, concomitant administration. n = p volunteers



Table 15.5.3 Individual concentrations table for metformin reference formulation, alone administration. n = p volunteers



PPD

Data about plasma concentration versus time for each subject, as well as the descriptive statistics are shown in tables 15.5.4 for gliclazide test formulation, 15.5.5 for metformin + gliclazide reference formulations concomitant administration and 15.5.6 for gliclazide reference alone administration.

Table 15.5.4. Individual concentrations table corresponding to metformin-gliclazide test formulation. n = P volunteers



Table 15.5.5 Individual concentrations table for metformin + gliclazide, reference formulation, concomitant administration. n = P volunteers



Table 15.5.6 Individual concentrations table for metformin reference formulation, alone administration. n = P volunteers

| | U-L- | | | | | | | | | | | Time | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Volunteer | 0.0000 | 0.5000 | 1,0000 | 20000 | 3.0000 | 4.0000 | 5.0000 | 6.0000 | 7.0000 | 8.0000 | 10.0000 | 120000 1 | 6.0000 2 | 24,0000 2 | 80000 3 | 2.0000 48.0 | 000 72.00 | 96,0000 | 120.0000 | 144,0000 168,000 | 00 |
| PPD | | | · | , | | | | | İ | | | | | | | | | | | | | |

PPD

Average values for the metformin and gliclazide's concentration obtained in the study as well as the descriptive statistics are shown in tables 15.5.7 and 15.5.8.

Table 15.5.7. Descriptive Statistics of the Values of the Metformin's Concentration in Biological Fluid

| | | | Metformin | -Giclazide | | | | 0 | abex <sup>®</sup> XR + C | iamicron MR | <b>#</b> | | | | Dabe | x <sup>®</sup> XR | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time | Mean | Median | Minimum<br>value | Maximum<br>value | Standar<br>deviation | CV% | Mean | Median | Minimum<br>value | Maximum<br>value | Standar<br>deviation | CV% | Mean | Median | Minimum<br>value | Maximum<br>value | Standar<br>deviation | CV% |
| PPD | ) | | 10.00 | Tulus | 00/000 | | | | 10.00 | Turus | ocrioton. | | | | Turus | 10105 | acriation. | |

Table 15.5.8 Descriptive Statistics of the Values of the Gliclazide's Concentration in Biological Fluid

| | | | Metformi | n-Glolazide | | | | 0 | abex®XR+[ | Diamicron MR | 1 | | | | Dabe | xª XR | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time | Mean | Median | Minimum<br>value | Maximum<br>value | Standar<br>deviation | CV% | Mean | Median | Minimum<br>value | Maximum<br>value | Standar<br>deviation | CV% | Mean | Median | Minimum<br>value | Maximum<br>value | Standar<br>deviation | CV% |
| PPD | | | 10.00 | TOTAL | acreson | | | | 10.00 | TOTAL | OCTIGLOII | | | | TOTAL | TOTAL | acriation | |

#### PPI

Figures 15.5.1 and 15.5.2 show the average charts in arithmetic and logarithmic scales, respectively, for gliclazide are shown in figures 15.5.3 and 15.5.4 in arithmetic and logarithmic scales.



Figure 15.5.1. Metformin's average concentration versus time chart in an arithmetic scale following the test and reference administration (standard deviation bars)



Figure 15.5.2. Metformin's average concentration versus time chart in logarithmic scale following the test and reference administration (standard deviation bars)



Figure 15.5.1. Metformin's average concentration versus time chart in an arithmetic scale following the test and reference administration (standard deviation bars)



Figure 15.5.2. Metformin's average concentration versus time chart in logarithmic scale following the test and reference administration (standard deviation bars)

#### 16. Estimation of Individual Pharmacokinetic Parameters

Non-compartmental computation of pharmacokinetic parameters was performed using the computer program Phoenix® WinNonlin® version 8.0 (PPD

The pharmacokinetic analysis was performed with a non-compartmental analysis, using real times following the dosing of the studied drugs. Pharmacokinetic parameters were determined as shown in tables 16.1. and 16.2, which include the individual values and descriptive statistics used for determining bioequivalence and drug-drug interaction, between the active ingredients, for metformin and gliclazide, respectively.

Table 16.1. Individual Data and Descriptive Statistics for Metformin's Pharmacokinetic Parameters ( $C_{max}$  in ng/mL,  $AUC_{0\rightarrow t}$  in h\*ng/mL and  $AUC_{0\rightarrow \infty}$  in h\*ng/mL).

| | Period | | C <sub>max</sub> | | | | | | | | AUC <sub>o.</sub> | | | | | | | AUC <sub>p</sub> a | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Volunteer | Form | Sequence | | Form | | A/B | Ln(A/B) | s/c | Ln(A/C) | | Form | | A/B | Lr(A/B) | A/C | Ln(A/C) | | Form | | A/B | Ln(A/B) | A/C | Ln(A/C) |
| | ABC | | A | В | ( | NO | u(A) | n/c | ui(r/c) | A | В | C | No | u(No) | n/c | ui(Ac) | A | 8 | C | - NO | ni(An) | n/c | LI(r)C) |
| PPD | i i | | | | | | | | | | | | | | | | | | | | | | |

Table 16.2. Individual Data and Descriptive Statistics for Gliclazide's Pharmacokinetic Parameters ( $C_{max}$  in ng/mL,  $AUC_{0\rightarrow t}$  in h\*ng/mL and  $AUC_{0\rightarrow \infty}$  in h\*ng/mL).

| | Period C <sub>ma</sub> | | | | | | AUC <sub>01</sub> | | | | | | | | ALC <sub>0.0</sub> | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Volunteer | | A | Form<br>B | С | A/B | Ln(A/B) | ĄC | Ln(A/C) | | Form<br>B | | A/B | Ln(A/B) | A/C | Ln(A/C) | | For B | , | A/B | Ln(A/B) | A/C | Ln(A/Q) |
| PPE | A B C | А | D | L | _ | | | | A | 0 | C | | | | | A | 0 | С | | | | |

The Phoenix WinNonlin NCA Core Output is provided in a separate listing.

# 17 Safety Evaluation

According to the Mexican Official Standard, NOM-177-SSA1-2013, there are several statistical tests to identify extreme values. Most of them start by calculating the student residual absolute value. Likewise, it is stated that "since studies are generally crossed designed, the most important extreme values is the extreme value for the subject".

An adequate method for estimating extreme values allows increasing reliability of the study conclusion. An analysis to identify outliers (extreme) values based on the student residual estimation among subjects will be performed using Bear software (current) for R environment.

Criterion: extreme values are those data which degree is higher than  $\pm$  2 standardized residuals intra-subject.

#### 17.1 Pharmacokinetic Parameters' Outliers

Outliers determination is by means of the intra-subject student residuals calculation according to the Mexican Official Standard, NOM-177-SSA1-2013; therefore, the potential outliers are those which exceed the criterion of  $\pm$  2 student residuals. In this study, outliers were determined according to Rasheed A. et al 2011, who states the statistical methodology to determine the outliers for the designs of more than two formulations, by means of the Andrew's curve. In figures 17.1.1, 17.1.2 and 17.1.3 the assessed pharmacokinetic parameters plots to determine the metformin's pharmacokinetic equivalence are shown, and in figures 17.1.4, 17.1.5 and 17.1.6 the assessed pharmacokinetic parameters plots to determine the gliclazide's pharmacokinetic equivalence are shown.

PPD

Figure 17.1.1. Intra-subject Student Residuals Plot for the Metformin's Pharmacokinetic Parameter Ln C<sub>max</sub>



Figure 17.1.2. Intra-subject Student Residuals Plot for the Metformin's Pharmacokinetic Parameter Ln AUC<sub>0-t</sub>



Figure 17.1.3. Intra-subject Student Residuals Plot for the Metformin's Pharmacokinetic Parameter Ln AUC<sub>0-∞</sub>



Figure 17.1.4. Intra-subject Student Residuals Plot for the Gliclazide's Pharmacokinetic Parameter Ln C<sub>max</sub>



Figure 17.1.5. Intra-subject Student Residuals Plot for the Gliclazide's Pharmacokinetic Parameter Ln AUC<sub>0-t</sub>



Figure 17.1.6. Intra-subject Student Residuals Plot for the Gliclazide's Pharmacokinetic Parameter Ln AUC₀-∞

#### 18. Adverse Events

All the information related with clinical results is included in clinical inform

#### 19 References

- Chow S.S, Liu JP. (2009). Design and Analysis of Bioavailability and Bioequivalence Studies. 3rd edition. US: CRC Press.
- Mexican Official Standard NOM-177-SSA1-2013 which sets out the tests and procedures
  to prove that a drug is interchangeable, requirements for the authorized third parties
  performing interchangeability tests; requirements for the conduct biocomparability studies,
  requirements for authorized third parties, research centers and hospitals conducting
  biocomparability tests.

#### 20 Appendices

- Quality Assurance Report.
- Individual Concentrations
- Winnonlin Core Outputs